CLINICAL TRIAL: NCT06500845
Title: Assessment of Marginal and Internal Fit of High Performance Polymer Endocrown Using Two Preparation Designs (Randomized Clinical Trial)
Brief Title: Assessment of Marginal and Internal Fit of High Performance Polymer PEEK Endocrown Using Two Preparation Designs
Acronym: PEEK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatema Khaled Mohammed Mansour, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 3324
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Endodontically Treated Molar; Marginal Fit; Internal Fit
Keywords: Endocrown

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and recruiters will not know the study group to which the next participant will be assigned.
  The trial participants, outcome assessors, and data analysis will be blinded after assignment to interventions.
  Emergency un-blinding: In cases of emergency to decrease or prevent any harms for the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Bevel marginal design endocrown for endodontically treated teeth
  Interventions: Other: Bevel marginal design endocrown for endodontically treated teeth
- Control group (Active Comparator): Butt marginal design endocrown for endodontically treated teeth
  Interventions: Other: Butt marginal design endocrown for endodontically treated teeth

INTERVENTIONS:
Other: Bevel marginal design endocrown for endodontically treated teeth — Bevel marginal design will be prepared for endodontically treated teeth and restores with Peek endocrown
  Arms: Intervention group
Other: Butt marginal design endocrown for endodontically treated teeth — Butt marginal design will be prepared for endodontically treated teeth and restores with Peek endocrown
  Arms: Control group

SUMMARY:
First, Participants in this study will be recruited according to inclusion criteria. Proper examination for the participants (clinically and radiographically). Preparation for endodontically treated molar for receiving high performance polymer endocrown. Checking and verification for the restoration (trying) and assessment of marginal and internal fit by replica technique. Then final cementation of endocrown.

DETAILED DESCRIPTION:
Examination and diagnosis:

Selection and examination of the patients according to inclusion and exclusion criteria. Diagnosis of the patient's chief complaint and teeth that will be involved in this study will be done.

Primary alginate impressions for diagnosis on primary casts and for mounting. The patients will be asked to maintain good oral hygiene measures by using tooth brush twice daily.

Taking a professional pre-operative photo.

Tooth preparation procedure:

Preparation of endocrown with two preparation designs on endodontically treated molars.

After tooth preparation, the final impression will be taken for each participant using polyvinyl siloxane impression and temporization of cavity using light curable temporary material.

Restoration trial appointment:

Endocrown try in and assessment of marginal and internal fit using replica technique with light body rubber impression.

Fabrication of final restoration:

Delivery of high performance polymer endocrown will be fabricated according to the two preparation designs; butt and bevel.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age range from 18 years -50 years old. They should be able to read and write so they can sign the informed consent.
2. Patient should have a good physical and psychologically state to be able to withstand the steps of the restoration procedure.
3. Have a molar with root canal filling with no active periodontal or apical involvement.
4. Patients having root canal treatment teeth indicated for endocrown treatment with 3 or 4 axial walls remaining.
5. Patient with axial wall length not less than 3 mm and not more than 5 mm.
6. Patient should have good oral hygiene and motivation.

Exclusion Criteria:

1. Patient with periodontal or apical involvement or improper root canal treatment.
2. Severe loss of the tooth structure in which the amount of the remaining tooth structure is less than 2mm.
3. Patient with poor oral hygiene or with occlusal instability
4. Patient with improper physical or psychological state.
5. Patient not pregnant or lactating.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-17 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Marginal fit | 2 weeks
  stereomicroscope by Micrometer

SECONDARY OUTCOMES:
Internal fit | 2 weeks
  stereomicroscope by Micrometer

CONTACTS AND LOCATIONS:
Overall Officials: Fatema K. Mansour, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No